CLINICAL TRIAL: NCT00954304
Title: Clinical Trial to Investigate the Duration of P-glycoprotein Inhibition After Oral Administration of HM30181AK Tablet in Healthy Male Subjects : An Open, Parallel Dose Group Design
Brief Title: Duration of P-glycoprotein Inhibition After Oral Administration of HM30181AK Tablet
Acronym: PGP inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Kyung-mi Park/ Director, Hanmi Pharmaceutical Company Limited
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-OXL-104
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Pgp inhibitor; P-glycoprotein inhibitor
MeSH Terms: interventions — Loperamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1mg group (Experimental): Administration of HM30181AK 1mg on day 4 and Loperamide 16mg (Loperamide 2mg x 8cap) on day 1,4,8,11,15
  Interventions: Drug: HM30181AK 1mg; Drug: Loperamide 2mg
- 5mg group (Experimental): Administration of HM30181AK 5mg on day 4 and Loperamide 16mg(Loperamide 2mg x 8cap) on day 1,4,8,11,15
  Interventions: Drug: HM30181AK 5mg; Drug: Loperamide 2mg
- 10mg group (Experimental): Administration of HM30181AK 10mg(HM30181AK 5mg x 2tab)on day 4 and Loperamide 16mg (Loperamide 2mg x 8cap) on day 1,4,8,11,15
  Interventions: Drug: HM30181AK 5mg; Drug: Loperamide 2mg
- 15mg group (Experimental): Administration of HM30181AK 15mg on day 4 and Loperamide 16mg (Loperamide 2mg x 8cap) on day 1,4,8,11,15
  Interventions: Drug: HM30181AK 15mg; Drug: Loperamide 2mg
- 60mg group (Experimental): Administration of HM30181AK 60mg on day 4 and Loperamide 16mg (Loperamide 2mg x 8cap) on day 1,4,8,11,15
  Interventions: Drug: HM30181AK 60mg; Drug: Loperamide 2mg

INTERVENTIONS:
Drug: HM30181AK 1mg — HM30181AK 1mg tablet
  Arms: 1mg group
Drug: HM30181AK 5mg — HM30181AK 5mg tablet
  Arms: 10mg group; 5mg group
Drug: HM30181AK 15mg — HM30181AK 15mg tablet
  Arms: 15mg group
Drug: HM30181AK 60mg — HM30181AK 60mg tablet
  Arms: 60mg group
Drug: Loperamide 2mg — Loperamide 2mg capsule

SUMMARY:
The purposes of this study are to investigate the duration of P-glycoprotein inhibition after oral administration of HM30181AK tablet in healthy male subject and proper dose of HM30181AK tablet.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers aged 20 to 50 years at screening
2. Subjects whose weights are heavier than or equal to 50 kg and ±20% of ideal body weight

   * Ideal body weight = (height cm - 100) x 0.9
3. Subjects who provided written, voluntary informed consent to participate in this clinical trial and to comply the directions including contraception after being fully informed of and understand this trial

Exclusion Criteria:

1. Subjects who have the clinically significant diseases or history in liver, kidney, nervous system, respiratory system, endocrine system, blood tumor and cardiovascular system.
2. History of the gastrointestinal diseases which may affect the absorption of oral drugs (e.g., Crohn's disease) or gastrointestinal operations (excluding simple typhlotomy and hernia repair).
3. The following results in laboratory test

   * AST, ALT > 1.25 x upper limits of normal
4. Systolic blood pressure below 100 mmHg or above 150 mmHg or diastolic blood pressure below 65 mmHg or above 95 mmHg in vital signs
5. History of drug allergy or other allergies which are clinically significant
6. History of drug abuse or positive reaction for drug abuse in urine screening test
7. Subjects who took prescription drugs or herbal medicines within 2 weeks prior to the first day of drug administration or OTC or vitamin preparations within 1 week prior to the first day of drug administration If the subjects meet other criteria, they could participate in the trial in the judgement of investigator.)
8. Subjects who have participated in other clinical trial within 2 months prior to the first day of drug administration
9. Whole blood donation within 2 months prior to the first day of drug administration or apheresis donation within 2 weeks prior to the first day of drug administration
10. Subject who are continuously drinking alcohol (over 21 units/week) or who cannot quit drinking during clinical trial period
11. Subject who are smoking over 10 cigar/day
12. Subjects who eat food containing caffeine or grapefruit or drink alcohol in prohibited period
13. Subjects who are inappropriate in the judgement of the investigator due to the reasons including clinical laboratory test results

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the duration of P-glycoprotein inhibition of HM30181AK by the Loperamide AUC measurement. | Day 1~Day 18

SECONDARY OUTCOMES:
Evaluate the PK parameters (Cmax, AUClast, AUCinf, Tmax, T1/2, CL/F etc) of HM30181AK by measuring the blood concentration of HM30181AK | Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea